CLINICAL TRIAL: NCT07256236
Title: A Single-arm, Multicenter, Phase II Study of Sacituzumab Tirumotecan (Sac-TMT/SKB264) in Combination With QL1706 for Recurrent or Metastatic Cervical Cancer
Brief Title: SKB264 Plus QL1706 in Recurrent or Metastatic Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHINE
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKB264+QL1706 (Experimental)
  Interventions: Drug: Sacituzumab tirumotecan; Drug: QL1706

INTERVENTIONS:
Drug: Sacituzumab tirumotecan — intravenous (IV) infusion (4mg/kg, Q2W)
  Other Names: SKB264; Sac-TMT; MK-2870
Drug: QL1706 — intravenous (IV) infusion (3mg/kg, Q2W). Continuous administration will be maintained until radiological disease progression, occurrence of intolerable toxicity, the participant requests to discontinue treatment, or other treatment discontinuation criteria specified in the protocol are met (whichever occurs first). The maximum duration of administration for QL1706 is 24 months.

SUMMARY:
This study is a prospective, single arm II clinical trial. The main objective of the study is to evaluate the efficacy and safety of the combination of Sacituzumab Tirumotecan (SKB264) and QL1706 in the treatment of recurrent or metastatic cervical cancer.

DETAILED DESCRIPTION:
Cervical cancer (CC) is a major global health concern. Current second-line options, including single-agent chemotherapy or PD-1/L1 inhibitors, provide limited benefit, with objective response rates (ORR) of only 5-29%. Patients with cervical adenocarcinoma, which constitutes 20-25% of cases, often have a poorer prognosis, and no specific treatments are recommended for this subtype.

QL1706, a novel dual anti-PD-1/CTLA-4 antibody, has been approved in China for the second-line treatment of CC. Separately, TROP2 is highly expressed in 88.7% of CC and is associated with poor prognosis. Sac-TMT, a TROP2-directed ADC, combined with an anti-PD-1 agent showed a promising ORR of 57.9% in a phase II study, without new safety signals.

Based on the unique mechanisms of action of Sac-TMT and QL1706, as well as the existing research data, their combination is expected to provide a better second-line treatment option for recurrent or metastatic CC. Therefore, we are applying to conduct this Phase II, multicenter, single-arm clinical study to evaluate the efficacy and safety of Sac-TMT in combination with QL1706 for the treatment of recurrent or metastatic CC, in order to improve clinical benefits for patients.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥18 years at the time of signing the informed consent form;
* Diagnosed with recurrent or metastatic cervical cancer [pathological types include squamous cell carcinoma, adenocarcinoma (excluding mucinous adenocarcinoma), and adenosquamous carcinoma, etc., with pathological report provided], and not suitable for radical treatments such as surgery or radiotherapy. Patients will be divided into the following two cohorts based on pathological type:

  * Cohort 1: Cervical squamous cell carcinoma;
  * Cohort 2: Cervical non-squamous carcinoma (including adenocarcinoma or adenosquamous carcinoma, and other types of cervical cancer)
* Have experienced failure of at least one prior line of platinum-based standard therapy or intolerance to platinum-based drugs in the recurrent or metastatic setting, or have experienced radiologically confirmed disease progression during or within 6 months after completion (≥4 cycles) of platinum-based neoadjuvant or adjuvant chemotherapy. Specific requirements are as follows:

  (a) Failure of first-line platinum-based standard therapy: meeting any one of the following criteria: i. Radiologically confirmed disease progression during treatment; ii. Radiologically confirmed disease progression after completion of treatment, provided the patient had a response (Complete Response (CR)/Partial Response (PR)/Stable Disease (SD)) and received ≥4 cycles of treatment; (b) Investigator's judgment that the subject is intolerant to platinum-based drugs; (c) Radiologically confirmed disease progression during or within 6 months after completion (≥4 cycles) of platinum-based neoadjuvant or adjuvant chemotherapy. Weekly chemotherapy administered concurrently with radiotherapy for sensitization purposes should not be counted as chemotherapy cycles;
* According to RECIST (v1.1) criteria, at least one measurable lesion (non-lymph node lesion with longest diameter ≥10 mm, or lymph node lesion with short diameter ≥15 mm). Lesions previously irradiated should not be selected as target lesions; unless there are no other measurable lesions available, in which case a previously irradiated measurable lesion that has shown confirmed progression radiologically may be selected as a target lesion. Subjects with only skin lesions or bone lesions are not eligible;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 within 7 days prior to dosing;
* Expected survival period ≥12 weeks;
* Subjects must have recovered from all toxicities resulting from prior therapy (i.e., improved to Grade 0 or 1, or to the level specified in the eligibility criteria), except for toxicities not considered a safety risk (such as alopecia, vitiligo, and other asymptomatic laboratory abnormalities). Subjects with ≤ Grade 2 neuropathy will be evaluated on a case-by-case basis in consultation with the investigator;
* Adequate organ and bone marrow function (without transfusion, recombinant human thrombopoietin, or colony-stimulating factor therapy within 2 weeks prior to dosing), defined as follows:

  1. Neutrophil count (NEUT#) ≥1.5×10⁹/L; Platelets (PLT) ≥100×10⁹/L; Hemoglobin ≥90 g/L;
  2. Liver function: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5 × ULN; for subjects with baseline liver metastases, ALT and AST ≤5 × ULN; Albumin ≥30 g/L; Total bilirubin (TBIL) ≤1.5 × ULN;
  3. Renal function: Creatinine clearance (Ccr) ≥50 ml/min (calculated using the standard Cockcroft-Gault formula); Urine protein ≤1+; if urine protein ≥2+, then 24-hour urine protein quantification must be ≤1.0 g;
  4. Coagulation function: International Normalized Ratio (INR), Activated Partial Thromboplastin Time (APTT), and Prothrombin Time (PT) ≤1.5 × ULN;
  5. Cardiac left ventricular ejection fraction (LVEF) ≥50%.
* For female subjects of childbearing potential, must agree to use effective medical contraception measures from the time of signing the informed consent form until 6 months after the last dose;
* The subject voluntarily joins this study, signs the informed consent form, and is able to comply with the visits and related procedures stipulated in the protocol.

Exclusion Criteria:

* Subjects who have had a known additional malignancy that is progressing or has required active treatment within the past 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, etc., that has undergone potentially curative therapy.
* Subjects with known leptomeningeal metastasis, brainstem metastasis, spinal cord metastasis and/or compression, or other active central nervous system (CNS) metastases. Subjects with brain metastases treated with local therapy may be enrolled if they meet the following criteria: clinically stable for at least 4 weeks, and no requirement for steroid treatment for at least 14 days prior to the first dose of study drug.
* Subjects with clinically significant cardiovascular diseases, such as: a) Presence of severe or uncontrolled cardiac disease or clinical symptoms requiring treatment within 6 months prior to the first study dose, including: congestive heart failure classified as New York Heart Association (NYHA) Class III or IV, unstable angina pectoris uncontrolled by medication, severe arrhythmia requiring drug treatment (except for atrial fibrillation or paroxysmal supraventricular tachycardia), and myocardial infarction; b) Previous history of myocarditis or cardiomyopathy; c) QTc interval > 480 ms based on baseline measurement.
* Subjects with severe and/or uncontrolled concurrent diseases, such as decompensated liver cirrhosis, nephrotic syndrome, uncontrolled hypertension or severe hypertension, clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Subjects diagnosed with active Hepatitis B or Hepatitis C.
* Subjects with known poorly controlled human immunodeficiency virus (HIV) infection, including HIV infection with a history of Kaposi's sarcoma and/or multicentric Castleman's disease.
* Subjects with known active tuberculosis.
* Subjects with a history of severe dry eye syndrome, meibomian gland dysfunction, blepharitis, or corneal diseases that affect timely corneal healing.
* Subjects with a known prior history of fistula of the female reproductive tract (e.g., vesicovaginal fistula, urethrovaginal fistula, vesicocervical fistula, etc.); subjects may be enrolled if the perforation or fistula has been treated with diversion surgery, resection, or repair, and the disease is considered by the investigator to have recovered or resolved.
* Subjects who have undergone major surgery (as defined by the investigator) within 30 days prior to the first dose of study treatment or have not recovered from prior surgery.
* Subjects with known allergy or hypersensitivity to the study drug or excipients; history of severe hypersensitivity to monoclonal antibodies.
* Subjects with a history of interstitial lung disease (ILD), or history of non-infectious pneumonitis requiring steroid treatment, or current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging during screening.
* Subjects with a history of allogeneic tissue/organ transplantation.
* Subjects with autoimmune disease that required systemic treatment within the past 2 years or requires immunosuppressive therapy during the study period. Subjects with controlled Type 1 diabetes, thyroiditis with normal thyroid function, hypothyroidism controlled well with hormone replacement therapy (HRT), or skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis) can be enrolled.
* Subjects who have previously received TROP2-targeted therapy, or any drug containing a topoisomerase I inhibitor, including antibody-drug conjugate (ADC) therapy.
* Subjects who have previously used any experimental anticancer vaccine, or any drug targeting T-cell co-stimulation pathways.
* Administration of a live vaccine within 30 days prior to the first dose of study treatment, or planned administration of a live vaccine during the study.
* Requirement for strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) within 2 weeks prior to the first dose of study treatment or during the study.
* Received any chemotherapy, radiotherapy, immunotherapy, or biologic therapy within 4 weeks prior to the first dose of study treatment; received small molecule tyrosine kinase inhibitors (TKIs), antitumor hormone therapy, systemic immunostimulants (including but not limited to interferon, IL-2), or Chinese herbal patent medicines with approved anti-tumor indications within 2 weeks prior to the first dose of study treatment.
* Received palliative radiotherapy to known metastatic sites within 2 weeks prior to the first dose of study treatment.
* Received systemic anti-infection therapy within 1 week prior to the first dose of study treatment.
* Any condition requiring systemic corticosteroid therapy (at doses >10 mg/day prednisolone or equivalent dose of similar drugs) or other immunosuppressive therapy within 14 days prior to the first dose of study treatment. However, subjects using intranasal, inhaled, topical, or local corticosteroid injections (e.g., intra-articular injection), or using corticosteroids as premedication for hypersensitivity reactions can be enrolled.
* Women who are pregnant or breastfeeding.
* Any condition that, in the investigator's judgment, interferes with the evaluation of the study drug, the subject's safety, or the interpretation of study results, or any other circumstance that the investigator considers inappropriate for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of patients who achieve complete response(CR) or partial response (PR), as assessed investigator per RECIST 1.1

SECONDARY OUTCOMES:
Overall Survival(OS) | From treatment administration up to a maximum duration of 24 months.
  Time from start of treatment to death due to any cause.
Progression Free Survival(PFS) | From treatment administration up to a maximum duration of 24 months.
  The time from the beginning of the patient's treatment to the disease progression per RECIST 1.1 based on investigator or death due to any cause, whichever occurs first.
Duration of Response(DoR) | Through study completion, an expected average of 24 months.
  DoR is defined as the time from the date of first documented CR or PR until date of documented disease progression per RECIST 1.1, as assessed by investigator or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | From treatment administration up to a maximum duration of 24 months.
  DCR is defined as the percentage of patients who achieve CR, PR or stable disease (SD), as assessed by investigator per RECIST 1.1
Percentage of Participants With Adverse Events (AEs) | Up to approximately 24 months.
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - First Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Affiliated Second Hospital, Fuzhou, Fujian
  - Zhangzhou Affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Second Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Qilu Hospital of Shandong University(Qingdao), Qingdao, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No